CLINICAL TRIAL: NCT01370928
Title: Colonoscopy Screening Using a Novel Slim Colonoscope - a Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PCF-Y0014-L
Record Dates: First submitted 2011-03-21; First posted 2011-06-10 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Colorectal Cancer; Adenomas
Keywords: Colonoscopy performance; Pain; Discomfort; Screening; Colorectal cancer; Colorectal cancer screening, diagnostics of adenomas
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prototype colonoscope (Experimental): The new colonoscope to be tested
  Interventions: Device: Olympus PCF-Y0014-L
- Standard colonoscope (Active Comparator): The standard colonoscope used world-wide today.
  Interventions: Device: Standard colonoscope

INTERVENTIONS:
Device: Olympus PCF-Y0014-L — Screening colonoscopy with a prototype colonoscope
  Other Names: Olympus PCF-Y0014-L colonoscope
  Arms: Prototype colonoscope
Device: Standard colonoscope — Screening colonoscopy
  Other Names: Olympus series 160 colonoscope
  Arms: Standard colonoscope

SUMMARY:
The purpose of this study is to compare the performance of a new prototype colonoscope with a standard colonoscope used world-wide today. The prototype colonoscope is more flaccid with a smaller diameter than the standard colonoscope. The hypothesis to be tested is that the prototype will improve negotiation of sharp bends and inflict less discomfort or pain to the patient. Both colonoscopes are manufactured by the same company.

ELIGIBILITY:
Inclusion Criteria:

* Persons included in the NordICC trial are eligible for inclusion
* For information about the NordICC trial see clinicaltrials.gov NCT00883792

Exclusion Criteria:

* Pregnancy
* Persons younger than 18 years
* Persons unable to comprehend the information given
* not possible to start the examination without prior administration of sedation/analgesics

Ages: 54 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Patients´ evaluation of pain and discomfort | 24 hours
  Analysis of validated feed-back questionnaires to be filled in on the day after the proceudre by the trial participants.

SECONDARY OUTCOMES:
Time used to reach the caecum | 1 hour
  The time used to reach the caecum will be recorded with a stop watch during the procedure.
Need for sedation/analgesics during the colonoscopy procedure | 1 hour
  If sedation/analgesics is administered during the colonoscopy procedure, the name of the agent, dose and route of administration will be recorded immediately.
Need to change to a different colonoscope to complete the procedure | 10 minutes
  If the colonoscopist decides to change to a different colonoscope during the procedure, the reason is recorded immediately after the procedure. The number of procedures where there is a change of colonoscope will be recorded.
Caecum intubation rate | 30 minutes
  The colonic segment reached during each colonoscopy is recorded immediately following the procedure. Caecal intubation rate describes the number of complete colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bretthauer, MD, Ph.d., Study Chair — Oslo University Hospital
Locations (1):
- Sørlandet Sykehus HF, Kristiansand, Norway

REFERENCES:
- [Derived] Garborg KK, Loberg M, Matre J, Holme O, Kalager M, Hoff G, Bretthauer M. Reduced pain during screening colonoscopy with an ultrathin colonoscope: a randomized controlled trial. Endoscopy. 2012 Aug;44(8):740-6. doi: 10.1055/s-0032-1309755. Epub 2012 May 23. PMID 22622786